CLINICAL TRIAL: NCT07017088
Title: A Randomized Crossover Trial on the Efficacy of Leuconostoc Mesenteroides (VITA-PB2) From Kimchi in Relieving Hangover Symptom
Brief Title: Efficacy of Leuconostoc Mesenteroides
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wonju Severance Christian Hospital (Other)
Responsible Party: Principal Investigator, Kyu Jae Lee, Prof., Wonju Severance Christian Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMB-2024-04
Record Dates: First submitted 2025-04-14; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Alcohol Drinking; Alcohol Drinking Related Problems
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Single group
  Treatment
  Interventions: Dietary Supplement: Leuconostoc mesenteroides

INTERVENTIONS:
Dietary Supplement: Leuconostoc mesenteroides — Control vs Experiment

SUMMARY:
Excessive alcohol intake can cause dehydration, digestive issues, oxidative stress, and hangover symptoms like headache and fatigue. Toxic metabolites like acetaldehyde and ROS contribute to liver damage. Chronic drinking activates harmful pathways like MEOS and increases inflammation. Gut-liver axis disruption also worsens hangovers. Probiotics, such as Leuconostoc mesenteroides, may help restore gut health and reduce toxicity, but more clinical research is needed.

ELIGIBILITY:
Inclusion

* Healthy adults aged between 30 and 60 years
* Body Mass Index (BMI) between 18.5 and 30 kg/m²
* Individuals with a history of hangover experience
* Adults with normal results in blood tests and vital signs
* No organic gastrointestinal disease found in endoscopy within the past 3 months
* Able to consume one bottle of soju within 30 minutes
* Individuals who have personally signed the informed consent form

Exclusion

* Individuals who have consumed excessive alcohol within the past week
* Individuals who participated in a human clinical trial within the past month
* Individuals taking supplements or medications that may affect alcohol metabolism
* Individuals with alcohol metabolism disorders, diabetes, hypertension, gallstones, pancreatitis, gout, active tuberculosis, gastrointestinal bleeding or surgery, or those with kidney, liver (e.g., hepatitis B/C carriers, alcoholic liver disease), heart, lung, gastrointestinal, or neurological diseases
* Pregnant women or those planning to become pregnant
* Individuals who have taken liver function supplements or similar medications/health products within one month before the study
* Individuals who consumed excessive alcohol within one week prior to study participation
* Any other individuals deemed unsuitable for the study by the principal investigator

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-08-13 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Assessment of Hangover Severity (Score, 0-10) Using the Alcohol Hangover Severity Scale (AHSS) | About 6 month
  Hangover severity will be assessed using the Alcohol Hangover Severity Scale (AHSS), a validated self-reported questionnaire that rates symptoms such as headache, nausea, fatigue, and dizziness on a 0-10 Likert scale. Higher scores indicate greater hangover severity, allowing for standardized comparison between groups.
Change in Blood Ethanol (mg/dL) and Acetaldehyde (mg/dL) Levels Over Time | 6 month
  Blood concentrations of ethanol and acetaldehyde (mg/dL) were assessed at multiple time points (0, 0.5, 1, 2, and 4 hours) following alcohol ingestion to evaluate the effect of VITA-PB2 supplementation on alcohol metabolism. This outcome measure helps determine potential differences in the metabolic clearance of ethanol and acetaldehyde between the intervention and placebo groups.
Change in Blood Aldehyde Dehydrogenase (ALDH) Activity (mU/mL) Over Time | 6 month
  Blood ALDH activity (mU/mL) was measured at 0, 0.5, 1, 2, and 4 hours following alcohol ingestion to evaluate the effect of VITA-PB2 supplementation on enzymatic metabolism of acetaldehyde. This outcome assesses potential group differences in ALDH activation as a marker of enhanced alcohol detoxification.

SECONDARY OUTCOMES:
Acute Hangover Scale (AHS) Total and Symptom-Specific Scores (0-7) After Alcohol Consumption | 6 month
  Hangover severity was evaluated using the Acute Hangover Scale (AHS), which assesses total and individual symptom scores (scale: 0 = none to 7 = incapacitating) across domains such as fatigue, headache, nausea, dizziness, and thirst. This measure was used to compare the impact of VITA-PB2 versus placebo on post-alcohol hangover symptoms.
Serum Liver Enzyme Levels-AST (U/L), ALT (U/L), and GGT (U/L)-for Safety Evaluation Post Alcohol Ingestion | About 6 month
  To evaluate the hepatic safety profile of VITA-PB2 supplementation, serum levels of liver enzymes-AST, ALT, and GGT (U/L)-were measured at 0, 0.5, and 4 hours after alcohol intake. This assessment helps determine any potential hepatotoxic effects or alterations in liver function associated with the intervention.
Plasma Reactive Oxygen Species (ROS; arbitrary units) and Nitrite (NO₂-; μM) Levels Following Alcohol Consumption | 6 month
  Plasma levels of reactive oxygen species (ROS) and nitrite (NO₂-), a stable metabolite reflecting nitric oxide (NO) production, were measured at multiple time points after alcohol ingestion to assess oxidative stress and NO signaling changes. This evaluation aimed to determine the antioxidant effects of VITA-PB2 supplementation in mitigating alcohol-induced oxidative damage.

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Kyu-Jae Lee, Wŏnju, Gangwon-do, South Korea

IPD SHARING:
Plan to Share IPD: No